CLINICAL TRIAL: NCT01369940
Title: NICHD Fetal Growth Study: Twin Gestations
Brief Title: The NICHD Fetal Growth Study: Twin Gestations
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911178; 11-CH-N178
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Fetal Growth Restriction; Growth Discordancy
Keywords: Growth Discordancy; Fetal Growth; Twin Growth
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NICHD Fetal Growth Study - Twin Gestations: Women with dichorionic twin gestations were enrolled between 8w0d and 13w6d and followed up to nine months (2012-2013) in this prospective cohort study.
  Intervention: No intervention

SUMMARY:
Normal growth and development of twins are important for the long-term health of the children. The purpose of this study was to empirically define the trajectory of fetal growth in dichorionic twins using longitudinal two-dimensional ultrasonography and to compare the fetal growth trajectories for dichorionic twins with those based on a growth standard developed by our group for singletons. This knowledge may lead to interventions that could minimize or prevent pregnancy and newborn health problems in the future.

DETAILED DESCRIPTION:
A prospective cohort of 171 women with twin gestations was recruited from eight U.S. sites from 2012 to 2013. After an initial sonogram at 11w0d-13w6d where dichorionicity was confirmed, women were randomized to one of two serial ultrasonology schedules. Ultrasound measurements at each follow-up visit included standard fetal biometrics ((BPD, HC, AC, FL); estimated fetal weight was calculated using a Hadlock formula. Growth curves and percentiles were estimated using linear mixed models with cubic splines. Percentiles were compared statistically at each gestational week between the twins and 1,731 singletons in the Fetal Growth Studies-Singletons cohort.

In addition to 2-D ultrasound measures for analyzing fetal growth, this study recorded maternal anthropometrics and a brief interview to capture changes in health status, stress and depression, and physical activity at each follow-up visit. Four blood draws at baseline and at targeted gestational ages for the eventual identification of biomarkers indicative of fetal growth were collected. After delivery, neonatal anthropometric measures were assessed for each twin, placental biospecimens were collected, and select information about the obstetrical course and newborn status were abstracted from medical charts. These exposures and outcomes provide opportunities to further compare singleton and twin gestations with respect to maternal biomarkers of fetal growth, well-being and maternal nutritional status using banked biospecimens to determine if the biomarkers ranges established for singletons are applicable to twin gestations.

Biospecimen Description:

* Maternal blood sample (serum, plasma, white blood cells, red blood cells and PAXgene RNA) at enrollment, 1st, 3rd, 5th follow-up visits, and delivery
* Cord blood and placentas for consenting women collected at delivery
* Placenta sample or buccal swab (determining zygosity by DNA probe for same sex pairs), collected at delivery

ELIGIBILITY:
INCLUSION CRITERIA:

* Twin, viable pregnancy
* 8+0 13+6 weeks of gestation
* Maternal age 18 - 45 years
* Spontaneous pregnancy or pregnancy from ovulation induction or in-vitro fertilization with known date of transfer
* Pregnancy from egg donor or embryo donor (record if anonymous or known source)
* LMP-date and crown-rump length measurement match within certain number of days according to a standard scheme (for larger twin)
* Expect to deliver at one of the participating hospitals

EXCLUSION CRITERIA:

* Fetal reduction (medically induced only)
* Congenital anomalies (structural or chromosomal)
* Either twin with an increased nuchal translucency (>99th percentile for crown-rump length; i.e. 3.5 mm or more)
* Monochorionic twins
* Crown-rump length discordancy >10% in dichorionic twin pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with dichorionic twin gestations, irrespective of the mode of conception, maternal medical history or obesity status, were enrolled from eight U.S. clinical centers. Women were enrolled between 8w0d and 13w6d, and accurate dating was required for enrollment. A total of 171 women were recruited, with 152 gestations resulting in live birth.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2011-05-29; Primary Completion 2013-08-25 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Fetal growth trajectories in dichorionic twin pregnancies | 3 years
  Fetal growth trajectories in dichorionic twin pregnancies were created using two- and selected three-dimensional ultrasound measures. Measures included maternal anthropometric measurements and 2D fetal biometry (BPD, HC, AC, FL) using standardized protocols.
  Women were recruited during the first trimester and followed until delivery. Each woman had seven scheduled ultrasound examinations, one at enrollment and six during follow-up visits. Women were randomized to receive sonograms according to one of the following two schedules: schedule A: 16, 20, 24, 28, 32 and 35 weeks or schedule B: 18, 22, 26, 30, 34 and 36 weeks.
Comparison of the fetal growth trajectories for dichorionic twins with singletons | 3 years
  The primary analysis compared fetal growth trajectories for dichorionic twins with 1,737 singleton gestations included in the NICHD Fetal Growth Studies - Singleton standard. For modeling twin trajectories, we used linear mixed models with a cubic spline mean structure and a random effects structure that included linear, quadratic, and cubic random effects for the twin pair and an intercept term for the individual fetus within twin pair. The linear mixed models were also used to test for overall differences (i.e., global tests) between the twin and singleton trajectories (for EFW and other measurements) using likelihood ratio tests of interaction terms between spline mean structure terms and twin-singleton indicator variables.
Incidence of fetal growth restriction (with small-for-gestational age as a proxy) in dichorionic twins (by zygosity) | 3 years
  Using small-for-gestational age as a proxy for growth restriction, we evaluated the percentage of dichorionic twins who would be classified below the 10th percentile using the study-generated singleton non-Hispanic white standard.
Comparison of singleton and twin gestations for maternal biomarkers of fetal growth | 3 years
  Longitudinal data will compare singleton and twin gestations with respect to maternal biomarkers of fetal growth, well-being and maternal nutritional status using banked biospecimens to determine if the biomarkers ranges established for singletons are applicable to twin gestations.

SECONDARY OUTCOMES:
Body composition | 3 years
  Pending the results of a validation study, measures of fetal fat and lean body mass from 2D ultrasound and/or fractional volumes from 3D will be assessed.
Genetic and environmental factors affecting fetal growth | 3 years
  Twin gestations offer an opportunity to differentiate genetic from environmental etiologies of developmental disorders, and to gain insight by investigating the role of shared factors versus factors affecting each of the twins independently. This involves comparing results of within cohort versus within twin pairs. The shared factors include maternal nutrition and gestational age, and the non-shared factors are those that affect each twin (e.g., placental placement, growth trajectory).
Biospecimen repository | 3 years
  The available bank of de-identified specimens will be used to add to our understanding of the determinants associated with fetal growth trajectories or adverse outcomes. The repository will be important for exploring possible epigenetic mechanisms and other specific hypotheses investigators may have.
Zygosity and growth trajectories | 3 years
  Placental samples for zygosity determination were obtained for all like-sex twin pairs. In the event that placental samples were not able to be obtained for like-sex twin pairs, a buccal swab from each infant was obtained prior to discharge, preferably in the first 48 hours of life. Both placenta zygosity samples and buccal swab samples were sent in real time to the Columbia Placenta Pathology Laboratory for zygosity testing. The research nurse provided women her with zygosity results when the information was available within three months following delivery.
Conception mode and growth trajectories | 3 years
  Information on mode of conception was collected during the enrollment interview.
Placental pathology and growth trajectories | 3 years
  The gross anatomy of the placentas (weight, cord length, diameter of the cord, and other gross morphology) were documented by the clinical site's participating pathologist. Photographs of placentas were taken by trained research personnel. Placental samples were obtained according to a standardized protocol. Eventual analysis may include proteomics, DNA analyses (e.g., comparative genomic hybridization, genomics, and assessment of the methylome), RNA expression, and microRNA levels. Also, analysis may include immunocytochemistry, histopathologic and biochemical / molecular studies. Once the research specimens were obtained, the remaining placenta was submitted to the clinical pathology department for processing and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Germaine M Louis, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University of California-Long Beach, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California
  - Christiana Care Health Services, Newark, Delaware
  - Northwestern University, Chicago, Illinois
  - National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland
  - Columbia University, New York, New York
  - Women and Infants, Providence, Rhode Island
  - Medical University of S. Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Grantz KL, Grewal J, Albert PS, Wapner R, D'Alton ME, Sciscione A, Grobman WA, Wing DA, Owen J, Newman RB, Chien EK, Gore-Langton RE, Kim S, Zhang C, Buck Louis GM, Hediger ML. Dichorionic twin trajectories: the NICHD Fetal Growth Studies. Am J Obstet Gynecol. 2016 Aug;215(2):221.e1-221.e16. doi: 10.1016/j.ajog.2016.04.044. Epub 2016 Apr 30. PMID 27143399
- [Derived] Amyx MM, Albert PS, Bever AM, Hinkle SN, Owen J, Grobman WA, Newman RB, Chien EK, Gore-Langton RE, Buck Louis GM, Grantz KL. Intrauterine growth discordance across gestation and birthweight discordance in dichorionic twins. Am J Obstet Gynecol. 2020 Feb;222(2):174.e1-174.e10. doi: 10.1016/j.ajog.2019.08.027. Epub 2019 Aug 24. PMID 31454510